CLINICAL TRIAL: NCT00004381
Title: Phase II Randomized Study of Tin Mesoporphyrin for Neonatal Hyperbilirubinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Rockefeller University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/12021; RUH-0330795A
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-10

CONDITIONS: Glucosephosphate Dehydrogenase Deficiency; Hyperbilirubinemia; Hemolytic Disease of Newborn
Keywords: glucose-6-phosphate dehydrogenase deficiency; hematologic disorders; hemolytic disease; hyperbilirubinemia; neonatal disorders; rare disease
MeSH Terms: conditions — Glucosephosphate Dehydrogenase Deficiency; Hyperbilirubinemia; Erythroblastosis, Fetal; Hematologic Diseases; Infant, Newborn, Diseases; Rare Diseases | interventions — tin mesoporphyrin

INTERVENTIONS:
Drug: tin mesoporphyrin

SUMMARY:
OBJECTIVES: I. Compare the efficacy of preventive vs. therapeutic tin mesoporphyrin in direct Coombs' test-positive ABO hemolytic disease of the newborn and glucose-6-phosphate dehydrogenase deficiency in infants living in Greece.

II. Assess the safety of tin mesoporphyrin in high-risk newborns.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients are stratified by gestational age and sex, and randomly assigned in pairs per stratum.

One group receives a preventive dose of tin mesoporphyrin. Another group receives a therapeutic dose of tin mesoporphyrin according to the plasma bilirubin concentration.

Patients in either group may be treated concurrently with phototherapy or exchange transfusion if clinically indicated.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Hyperbilirubinemia associated with either of the following: Direct Coombs' test-positive ABO hemolytic disease of the newborn Glucose-6-phosphate dehydrogenase deficiency --Prior/Concurrent Therapy-- No maternal phenobarbital in last month of pregnancy --Patient Characteristics-- Performance status: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: No congenital renal abnormality Cardiovascular: No congenital heart abnormality Pulmonary: No asphyxia requiring assisted ventilation at delivery Other: Gestational age more than 210 days Birth weight at least 1500 g No other major congenital abnormality, i.e.: Central nervous system Chromosomal Gastrointestinal No evident or suspected congenital infection, e.g.: Cytomegalovirus Herpes Rubella Syphilis

Ages: 0 Years to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1999-12

CONTACTS AND LOCATIONS:
Overall Officials: Attallah Kappas, Study Chair — Rockefeller University
Locations (2):
- United States (2):
  - New England Medical Center Hospital, Boston, Massachusetts
  - Rockefeller University Hospital, New York, New York